CLINICAL TRIAL: NCT02565901
Title: A Phase 1-2 Study of Sirolimus, Docetaxel and Carboplatin for Treatment of Patients With Metastatic, Castration Resistant Prostate Cancer: (Rapamycin Inhibition of DDSP [RID])
Brief Title: Sirolimus, Docetaxel, and Carboplatin in Treating Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to insufficient funding
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bruce Montgomery, Professor, Medical Oncology Division University of Washington School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9388; NCI-2015-01478 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9388 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); P50CA097186 (NIH); RG1715104 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2015-09-25; First posted 2015-10-01 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer AJCC v7; Metastatic Malignant Neoplasm in the Bone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Docetaxel; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (sirolimus, docetaxel, carboplatin) (Experimental): Patients receive docetaxel IV over 30-60 minutes and carboplatin IV over 30 minutes on day 1. Beginning in cycle 2 and continuing in subsequent cycles, patients also receive sirolimus PO on day -2. Treatment repeats every 21 days for 10 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Sirolimus
- Arm II (sirolimus, docetaxel, carboplatin) (Experimental): Patients receive sirolimus PO on day -2. Patients also receive docetaxel IV over 30-60 minutes and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 10 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Sirolimus

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217

SUMMARY:
This partially randomized phase I/II trial studies the side effects and how well sirolimus works when given together with docetaxel and carboplatin in treating patients with castration-resistant prostate cancer that has spread to other places in the body (metastatic). Biological therapies, such as sirolimus, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving sirolimus together with docetaxel and carboplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the recommended phase 2 dose (RP2D) of sirolimus combined with docetaxel and carboplatin in the treatment of metastatic castration resistant prostate cancer (CRPC). (Phase I)

II. To assess the effectiveness of sirolimus in suppressing the induction of the deoxyribonucleic acid (DNA) damage secretory component WNT16B in tumor stroma following docetaxel and carboplatin. (Phase II)

EXPLORATORY OBJECTIVES:

I. To assess maximal prostate-specific antigen (PSA) response to sirolimus combined with docetaxel and carboplatin. (Phase I)

II. To assess PSA response duration to sirolimus combined with docetaxel and carboplatin. (Phase I)

III. To assess response of measurable disease. (Phase I)

IV. To assess time to progression of bone lesions or measurable disease (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1). (Phase I)

V. To assess effect of sirolimus with docetaxel and carboplatin on DNA damage surrogates in cancer associated stroma compared to untreated and docetaxel and carboplatin treated stroma. (Phase I)

VI. To assess maximal PSA response to sirolimus combined with docetaxel and carboplatin. (Phase II)

VII. To assess PSA response duration to sirolimus combined with docetaxel and carboplatin. (Phase II)

VIII. To assess response of measurable disease (RECIST 1.1). (Phase II)

IX. To assess time to progression of bone lesions or measurable disease (RECIST 1.1). (Phase II)

X. To assess toxicity of the RP2D dose of sirolimus with docetaxel and carboplatin. (Phase II)

XI. To determine the effect of docetaxel and carboplatin therapy on the DNA damage secretory program (DDSP) in serum. (Phase II)

XII. To determine response to sirolimus, docetaxel and carboplatin in tumors with mutation of DNA repair pathway genes (breast cancer gene 2 [BRCA2], ataxia telangiectasia mutated [ATM] and other Fanconi anemia complementation groups [FANC] pathway members). (Phase II)

XIII. To correlate the presence of DNA repair pathway mutations in circulating tumor cells (CTC) and circulating tumor DNA (ctDNA) with tumor biopsy and correlate changes in CTC number and ctDNA mutation levels with clinical responses. (Phase II)

OUTLINE: This is a phase I, dose de-escalation study of sirolimus followed by a phase II study.

PHASE I: Patients receive sirolimus orally (PO) on day -2*. Patients also receive docetaxel intravenously (IV) over 30-60 minutes and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 10 cycles in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive docetaxel IV over 30-60 minutes and carboplatin IV over 30 minutes on day 1. Beginning in cycle 2 and continuing in subsequent cycles, patients also receive sirolimus PO on day -2. Treatment repeats every 21 days for 10 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive sirolimus PO on day -2. Patients also receive docetaxel IV over 30-60 minutes and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 10 cycles in the absence of disease progression or unacceptable toxicity.

* NOTE: Patients receive sirolimus 2 days prior to chemotherapy day 1 (there is no day 0).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) providing agreement to adhere to the dosing schedule, report for all trial visits and authorization, use and release of health and research trial information
* Histologically or cytologically confirmed carcinoma of the prostate (excluding neuroendocrine differentiation or squamous cell histology)
* Ongoing gonadal androgen deprivation therapy with gonadotropin-releasing hormone (GnRH) analogues, antagonists or orchiectomy; patients who have not had an orchiectomy must be maintained on effective GnRH analogue/antagonist therapy
* Castration resistant prostate cancer as defined by serum testosterone < 50 ng/ml and at least one of the following:

  * PSA level of at least 2 ng/ml that has risen on at least 2 successive occasions at least 1 week apart
  * Evaluable disease progression by modified RECIST 1.1
  * Progression of metastatic bone disease on bone scan with > 2 new lesions
* Prior therapy with abiraterone, enzalutamide and/or docetaxel; if a patient has not received docetaxel or cabazitaxel chemotherapy, the patient must be informed of this treatment choice as an alternative; if the patient has received docetaxel or cabazitaxel chemotherapy or refuses one of both of these therapies, this rationale must be documented and the patient is then eligible; patient must be offered and made aware of all Food and Drug Administration (FDA)-approved treatment options; patients with bone only disease may not have received radium-223
* The presence of metastatic disease amenable to computed tomography (CT) or ultrasound guided biopsy; this may include thoracolumbar vertebral bodies, pelvis, femur or humerus or soft tissue or nodal metastasis amenable to biopsy (excluding lung or pleural lesions)
* Agree to participate in biopsy of metastatic lesion during the study at day 21
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Life expectancy >= 12 weeks
* No prior malignancy is allowed except:

  * Adequately treated basal cell or squamous cell skin cancer or
  * In situ carcinoma of any site or
  * Other adequately treated malignancy for which the patient is currently disease free for at least one year
* Patients with any prior chemotherapy regimens are eligible
* Patients with disease only in the bone may not have received Xofigo/radium 223 to avoid ongoing DNA damage in bone marrow
* Patients who are or are not receiving bisphosphonates or denosumab are eligible; bisphosphonates or denosumab should not be initiated after registration and during active treatment
* Absolute neutrophil count >= 1.5 x 10^9 cells/L (within 14 days prior to registration)
* Hemoglobin (Hgb) >= 9.0 g/dL (within 14 days prior to registration)
* Platelets >= 100,000 x 10^9/L (within 14 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 x upper limit of normal (ULN) (within 14 days prior to registration)
* Total bilirubin =< 1.5 x ULN (within 14 days prior to registration)
* Serum creatinine < 1.5 X institutional ULN mg/dL OR estimated glomerular filtration rate (eGFR) >= 50 mL/min (within 14 days prior to registration)

Exclusion Criteria:

* Patients currently receiving active therapy for other neoplastic disorders
* Patients with histologic evidence of small cell carcinoma of the prostate will not be eligible
* Patients with disease only in the bone previously treated with radium-223 will not be eligible
* Known parenchymal brain metastasis
* Active or symptomatic viral hepatitis or chronic liver disease
* Estimated creatinine clearance less than 50 ml/minute
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) class II-IV heart disease
* Atrial fibrillation, or other cardiac arrhythmia requiring medical therapy
* Administration of an investigational therapeutic within 30 days of cycle 1, day -2
* Patients with dementia/psychiatric illness/social situations that would limit compliance with study requirements or would prohibit the understanding and/or giving of informed consent
* Patients with medical conditions, which, in the opinion of the investigators, would jeopardize either the patient or the integrity of the data obtained will not be eligible
* Any condition which, in the opinion of the investigator, would preclude participation in this trial
* Patients on anticoagulation therapy which cannot be held for metastatic biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montgomery, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Group: Patients treated with docetaxel, carboplatin and sirolimus in the phase 1 component of study
Period: Overall Study
Arm/Group | Arm I (Sirolimus, Docetaxel, Carboplatin) | Arm II (Sirolimus, Docetaxel, Carboplatin) | Phase 1 Group
Started | 11 | 11 | 6
Completed | 11 | 11 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Sirolimus, Docetaxel, Carboplatin) | Arm II (Sirolimus, Docetaxel, Carboplatin) | Phase 1 Group | Total
Number analyzed (Participants) | 11 | 11 | 6 | 28
Age, Continuous [Median (Full Range); unit: years] | 72 [68 to 82] | 75 [68 to 82] | 73 [68 to 82] | 72 [68 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 11 | 11 | 6 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 11 | 5 | 26
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1
  White | 11 | 8 | 5 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 6 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Deoxyribonucleic Acid (DNA) Damage Secretory Program Induction (DDSP) (Phase II)
Description: Will be determined by the level of genetic expression of WNT16, IL6, or SFRP2 in tissue after chemotherapy (carboplatin/docetaxel) compared to background/baseline measurement. The primary metric of DDSP induction will be quantitative reverse transcription-polymerase chain reaction, which is quantitative, but in the event of ribonucleic acid degradation in sample processing, the alternative measure will be immunohistochemistry (0-2 scale of expression).
Time Frame: Baseline up to day 21 after starting treatment
Population: Results do not exist. Because of COVID, the laboratory which would have performed the analysis was shut down for an entire year and inadequate funding exists for data analysis.
Groups:
- Arm I (Sirolimus, Docetaxel, Carboplatin): Patients receive docetaxel IV over 30-60 minutes and carboplatin IV over 30 minutes on day 1. Beginning in cycle 2 and continuing in subsequent cycles, patients also receive sirolimus PO on day -2. Treatment repeats every 21 days for 10 cycles in the absence of disease progression or unacceptable toxicity.
  Carboplatin: Given IV Docetaxel: Given IV Laboratory Biomarker Analysis: Correlative studies Sirolimus: Given PO
Arm/Group | Arm I (Sirolimus, Docetaxel, Carboplatin) | Arm II (Sirolimus, Docetaxel, Carboplatin)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Incidence of Adverse Events Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (Phases I and II)
Description: Safety will be assessed through summaries of adverse events, vital signs, physical examinations, and clinical laboratory test data. Adverse events will then be quantified via CTCAE 4.0.
Time Frame: Up to 3 years
Measure: Number; unit: Grade 3 or 4 AE
Arm/Group | Arm I (Sirolimus, Docetaxel, Carboplatin) | Arm II (Sirolimus, Docetaxel, Carboplatin) | Phase 1 Group
Number analyzed (Participants) | 11 | 11 | 6
Grade 3 or 4 AE | 2 | 2 | 0

3. Secondary Outcome: Percentage of Patients With Reduction in Prostate Specific Antigen According to the Prostate Cancer Working Group 2 (PCWG2) Criteria (Phases I and II)
Description: PSA decline from the level at registration will be quantified for each patient and proportion of patients with PSA decline divided by the total number of patients enrolled in study will be described.
Time Frame: Baseline to up to 3 years
Measure: Number; unit: Percent with PSA decline
Arm/Group | Arm I (Sirolimus, Docetaxel, Carboplatin) | Arm II (Sirolimus, Docetaxel, Carboplatin) | Phase 1 Group
Number analyzed (Participants) | 11 | 11 | 6
Percent with PSA decline | 36 | 36 | 50

ADVERSE EVENTS:
Time Frame: During time on study to 30 days after last therapy. This was up to 2 years.
Description: CTCAE 4.0 definitions of adverse events were used. Patients were evaluated with complete blood counts and comprehensive panels with each cycle and as clinically indicated
Arm/Group | Arm I (Sirolimus, Docetaxel, Carboplatin) | Arm II (Sirolimus, Docetaxel, Carboplatin) | Phase 1 Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 2/11 | 2/11 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Sirolimus, Docetaxel, Carboplatin) (N=11) | Arm II (Sirolimus, Docetaxel, Carboplatin) (N=11) | Phase 1 Group (N=6)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) — Grade 3 or greater neutropenia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT02565901/Prot_SAP_000.pdf